CLINICAL TRIAL: NCT06844331
Title: ULtrasOund Applicability in the Assessment of Patients With fibRosing Interstitial Lung Disease (LORD): A Research Protocol of a Single Center, Real-life, Prospective Observational Study
Brief Title: Ultrasound Applicability in the Assessment of Patients With Fibrosing Interstitial Lung Disease
Acronym: LORD
Status: Enrolling by invitation | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S-20220036
Record Dates: First submitted 2025-02-14; First posted 2025-02-25 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Fibrosing Interstitial Lung Diseases; Thoracic Ultrasound
Keywords: Fibrosing interstitial lung diseases; Thoracic ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- F-ILD patients: The investigators including the patients with fibrosing interstitial lunge disease (F-ILD) as cohort.
  Both the patients with idiopathic interstitial lung diseases and progressive pulmnoary fibrosis will include.
  Interventions: Device: Thoracic ultrasound

INTERVENTIONS:
Device: Thoracic ultrasound — The investigators want to investigate that TUS/US can use to identify and to monitir the disease progression in the patients with F-ILD
  Other Names: Ultrasound

SUMMARY:
In this study the investigators want to examine the different ultrasound techniques to assess the patients with lung fibrosis.

The investigators want to followup these patients in 1 year to see the changes in lungs, pleura, diaphragm and measurments of overarm and thigh muscles to see that the investigators can identify the patients with lung fibrosis with this methods and monitor the progression.

Now a days the CT scan in the lungs needs to monitor these participants, but the investigators want to see the ultrasound can use insted for CT scanning to minitor these pateints.

These patient group has very bad prognosis, so it is necessary to identify these patients as early as possible to treatments.

DETAILED DESCRIPTION:
Introduction Fibrosing interstitial lung diseases (F-ILD) represent a heterogeneous disease category involving many subtypes with different clinical, radiological and histological characteristics . Idiopathic pulmonary fibrosis (IPF) is the most common subtype of F-ILD, and IPF is the prototype of other F-ILD phenotypes, known as progressive pulmonary fibrosis (PPF). Despite their diverse presentation, the common denominator defining them as F-ILD patients is due to similarities regarding irreversible symptom worsening, decline in lung physiological parameters and progression of pulmonary fibrosis on thoracic imaging . Accomplishment of early F-ILD diagnosis and disease progression is crucial to initiate treatment at early stage of disease. Chest high-resolution computed tomography (HRCT) is considered the golden standard to diagnose and quantify pulmonary fibrosis. However, repeated HRCT performance is time-consuming, and repeated HRCT scanning is hampered by the cumulated radiation exposure with the increasing risk of cancer development.

Therefore, it is necessary to propose new modalities for the early identification and monitoring of disease progression in F-ILD patients.

Thoracic ultrasound (TUS) is superior to diagnose various conditions of the lung parenchyma and pleura compared to chest X-ray (CXR) . B-line artefacts (BLA) and the interstitial syndrome (IS) are well described TUS indicators related to ILD, and several studies have described a linear correlation between an increasing number of BLAs and the severity degree of fibrotic HRCT findings based on a Warrick score . Additionally, a significant negative correlation between an increased distance between BLAs and decreasing lung physiological parameters has also been demonstrated. Not only parenchymal, but also pleural abnormalities (PA) occur in patients with F-ILD. Several studies have proposed that increasing thickness and irregularity of the pleura can be used as a tool to assess disease severity in patients with F-ILD.

Less investigated ultrasound (US) modalities within F-ILD are diaphragm excursion (DE) and lung ultrasound share wave elastography (LUSWE). Different methods have been used to evaluate DE . According to current evidence, IPF patients were found to have a lower DE compared to healthy individuals, and restrictive ventilation pattern with lower values of forced vital capacity (FVC) was also associated with lower DE . These findings may be explained by a combination of lung compliance reduction ("lung stiffness") and development of diaphragm muscle atrophy over time in patients presenting with F-ILD traits where further development of hypoxemia and immobilization in severe disease stages may develop to sarcopenia.

LUSWE is based on measuring the velocity of the US waves' propagation along the lung surface from a given surface point (intercostal space), where the velocity is dependent on the change in wave phase with distance. The velocity of the US waves increases with tissue stiffness as consequence of reduced elastic properties. In two observational studies distinct higher LUSWE velocities were found in ILD patients compared to healthy individuals, and furthermore a negative correlation between LUSWE velocities and FVC and interstitial lung abnormalities was observed . Therefore, LUSWE may be a valuable supplementary and clinical tool not only to identify F-ILD but also to separate F-ILD from non-fibrotic ILD.

As previously described patients with F-ILD will in addition to increased dyspnea over time, also develop weight loss due to sarcopenia. Sarcopenia is defined as loss of muscle strength, endurance (muscle quality), and muscle mass (muscle quantity), and part of the frailty syndrome defined by a combined loss of functional reserves across different domains (e.g. physical ability, cognition, and energy) resulting in negative implications on health status in multimorbid and especially older patients . The European Working Group on Sarcopenia in Older People 2 (EWGSOP-2) has established diagnostic consensus criteria in which the diagnosis of sarcopenia is made by assessing 1) physical function either by chair stand test or hand-grip strength, by hand dynamometer and 2) estimating the appendicular lean mass. The latter can be done by using B-mode US and anthropometric measurements the appendicular lean mass (ALM) can be estimated. The established thresholds for ALM for men and women have been defined (<20 kg and <7, 0 kg/m2 for men and <15 kg and < 5,5kg/m2 for women).

The main challenge in comparing study results on TUS/US in patients with F-ILD is the heterogeneity in the methodology with use of different TUS/US protocols in incomparable cohorts with a mixture of different ILD subtypes, where some subtypes present with a more fibrotic pattern than others. In this context, it is problematic to determine the diagnostic value of TUS/US for a specific F-ILD category. Some studies have investigated on TUS use in patients with IPF , but most of the studies on patients with F-ILD are of observational nature with cross-sectional designs and primarily performed in patients with underlying autoimmune rheumatic diseases . At present, no studies have accomplished real-life prospective TUS/US follow-up, including promptly investigated TUS/US modalities such as BLA, IS, and PA, and less investigated TUS/US modalities such as DE, LUSWE and ALM, and dealt with these TUS/US modalities as a monitoring tool for F-ILD disease activity or treatment response, and is thus an area encumbered with a significant knowledge gap. The latter was emphasized in the recent European Respiratory Society statement on TUS that warrants studies assessing the impact of these points as areas of future TUS/US research .

Hypotheses The investigators hypothesize that TUS/US modalities such as BLA, IS, PA, DE, LUSWE, and ALM are clinically valuable, both individually and in combination for identifying F-ILD and monitoring disease activity. These modalities are expected to correlate with FVC, diffusion capacity of the lung for carbon monoxide (DLCO), HRCT findings, and clinical symptoms. In such, F-ILD patients with severe disease are hypothesized to present with TUS/US findings as increased number of BLAs, increased pleura thickness with irregularity, decreased DE, higher LUSWE velocities, and lower ALM values. Furthermore, these parameters are proposed to serve as dynamic indicators of F-ILD disease activity over time.

Statistical analyses To assess the reproducibility of our sample the investigators conducted descriptive statistics. Categorical outcomes were presented as numbers and percentages and non-categorical outcomes were presented as either median and interquartile range or mean and standard deviation, depending on the normality of the variable.

The primary objective where to evaluate the predictive value of the longitudinal measured TUS/US modalities on the outcomes HRCT, Warrick score and its subscales, PFT, 6MWT and PROMs. Hence the investigators utilize a mixed effect model including a random intercept. The evaluation of the model predictive performance will be assessed by way of reliability (including intra and inter rater reliability) based on the intra class correlation coefficient and agreement evaluated by Bland-Altman plots with 95% limits of agreement. The discrepancy will be defined as the difference between the predictive and true value of the outcome based on the mixed effect model.

For sensitivity purposes the investigators will also assess the predictive of specific characteristics of HRCT by way of descriptive statistics.

Missing data will be assumed to be missing either completely at random or at random, and thus will handled implicitly by maximum likelihood estimation.

All analyses will be performed using either Stata SE 16.1 (StataCorp, College Station, TX, USA) or the statistical software R, 95% confidence intervals will be reported and a p-value less than 0.05 will be considered statistically significant.

Ethics The study will be conducted in accordance with the Declaration of Helsinki with written patient consent of included patients after prior oral and written project information. The patient can withdraw her/his statement of commitment at any time. The law on the processing of personally identifiable information will be complied with and data from the project will be stored in accordance with Odense University Hospital's guidelines. The project is approved by the Danish Data Protection Agency (Ref. no. 22/45135) and the Science Ethics Committee for the Region of Southern Denmark (Ref. no. S-20220036).

Patient recruitment Respiratory physicians from SCILS, Department of Respiratory Medicine at Odense University Hospital will recruit patients who prior to follow-up in SCILS have received recruitment material. Patients, who are willing to participate in LORD study will be contacted by the PhD student, where an agreement for information and obtainment of detailed oral and written consent will be planned. This meeting will take place in the outpatient clinic of SCILS under quiet circumstances, and the patient will be given 24 hours to consider participation. The patients who are willing to participate will be included after obtain their oral and written consent. Other patients, who are not willing to participate will follow up in the rutine SCILS clinic.

HRCT A standard HRCT scan with inspiratory and expiratory image sections on average results in the patient having a radiation dose of approx. 6-7 mSv (Sievert definition: SI unit for the dosage of ionizing radiation equal to 100 rems. 1 Sv = 1 Sievert = 100 rem = 1 J/kg ((this is based on calculations from The National Institute of Radiation Hygiene (Danish: "Statens Institut for Strålehygiejne")). It is theoretically calculated that such a radiation dose entails a risk of developing cancer of 0.01-0.1%, meaning that the total lifetime risk of developing a cancer disease increases from 25% (which applies to the entire population) to 25.1%. In this population of patients this risk is considered negligible.

TUS/US In TUS/US examinations, sound waves are converted into images on a TV screen. No side effects have been reported with the use of US. Apart from a slight pressure experienced when the ultrasound head touches the chest, the US examination is painless with minimal discomfort for the patient (37). As there are no immediate disadvantages or risks associated with TUS/US, the study only seems to contribute with advantages in form of clinically relevant information.

Sample size The endpoint used for sample size calculation is the ability of TUS performed at 12 months follow-up to detect disease progression using HRCT findings at 12 months as the golden standard. With an expected overall prevalence of the F-ILD phenotype of 14-32% among patients with ILD(38, 39), significance level of 0.05, power of 80%, an expected TUS sensitivity of 70-80%, and assuming the clinical use of US would be as a screening test prior to HRCT confirmation, the calculated sample size is estimated to be between 31 (sensitivity 70%) and 107 patients (sensitivity 80%) (40). Patients with F-ILD are associated with increased mortality, why some patients will not be alive at 12 months follow-up. A conservative estimate is that 10% of the patients will not complete or have died within the 1-year follow-up following inclusion. Adjusting for a 10% drop-out at 12 months follow-up will increase the total sample size to be between 34 and 117 patients with F-ILD. Since the study is performed as part of a PhD programme and 12 months follow up time is needed, the inclusion period necessities to be restricted to 12 months to ensure feasibility within the three year time frame of the PhD programme. Based on the sample-size calculations and the inclusion period restrictions the study will aim to include up to 117 patients or as many as possible with at least 34 patients within the inclusion period of 12 months.

Patient involvement Our study will actively involve patients and their relatives in all aspects of the research process which involves that protocol details, recruitment material and information documents have presented and been discussed with patients in our clinic prior to their final editions. The project group consider it essential to include patients as early in the research process as possible to adjust their needs and experiences, which may have crucial impact on how the projects are being planned. The project group responsible for this project in SCILS at the Department of Respiratory Medicine will orally inform the relevant group of potential patients about the project and provide written information materials. Written consent will be obtained prior to inclusion.

Discussion The LORD study is a single-center, real life, prospective observational study examining patients with F-ILD three times over a follow-up period of 12 months according to whether several different US modalities (BLA, IS, PA, DE with area-method and M-mode, LUSWE and ALM) can be used to diagnose and identify disease progression. To the best of our knowledge, this is the first study to explore multiple TUS/US modalities within this patient category in a longitudinal set-up.

The investigatrs plan to examine not only most conventional investigated TUS modalities such as BLA and PA , but also less investigated US modalities such as LUSWE and diaphragm excrusion on basis of the above mentioned methods. Additionally, the ALM modality has the potential to monitor changes in muscle quality and quantity over time in these often fragile patients, an area that has not been thoroughly investigated in patients with F-ILD.

Thought TUS/US has been increasingly used in the past two decades, the overall evidence in this area is heterogeneous in nature, both regarding to F-ILD subtypes but also applied TUS/US protocols . Therefore, our study intend to clarify a detailed and enhanced perspective on the application of TUS/US modalities in patients with F-ILD, both single but also composite for identification of diagnosis and disease progression.

The diagnostic delay of F-ILD is considerable high approximating two years, and further the mortality rate is high in this patient group compared to other chronic lung diseases. Up to now no curative medicine have been found for F-ILD, but two antifibrotic therapies are available, Pirfenidon and Nintedanib, which delay the disease progression and in such indirectly increases survival. This emphasizes the importance of early detection and prompt treatment initiation in patients with F-ILD, why the investigators await our results in anticipation.

Several strengths and limitations should be addressed:

TUS has already described as a relevant screening modality in other F-ILD and with other US modalities (LUSWE, DE and ALM) it can use to screen patients with F-ILD in a better and promising way. Our study aims to show that TUS/US modalities is feasible and useful method that can use to monitor and early detect disease activity in F-ILD patients.

TUS/US are radiation free modalities that can performed in same day of consultation, and it is easily accessible.

Patients that are included in our study are assessed in MDT conferences in tertiary ILD center in Denmark, and it reduced the selection bias and false classification on diagnosis (information bias) as well as a homogeneous group of F-ILD.

The investigators planned to follow-up patients in baseline, after 180 and 365 days performing PFT, 6MWT, clinical examination and TUS/US on same day.

All the TUS/US findings validated HRCT as golden standard, and HRCT examined by a subspecialized HRCT radiologist , who is blinded from clinical, paraclinical and TUS/US data. It gives low intraobserver variability to our study.

The PhD student perform TUS/US scanning to all the included patients. It also gives low intraobserver variability.

The main limitation in our study is that unable to carry out the HRCT scanning and TUS/US in same day. According to hospital setup in Denmark, it is not possible to carry out HRCT in same day with TUS/US. This may interferer the correlation between HRCT and ultrasound. However, PFT, 6MWT, clinical examination and US examination will conducted in same day.

HRCT is performing in several centers can also be a limitation. The patients referred to our center from the peripheral hospitals with HRCT scanning. There can be differences in scan machines, setup and scanning protocols. However, as mentioned earlier all the HRCT scanning assessed by the subspecialized HRCT radiologist who is blinded from US results and other data.

Our study is a single center study and not 100% generalized to other F-ILD cohorts. There can be an intrainstitutional bias.

Furthermore, performing several different TUS/US modalities require training, can be examiner dependent, and there are 3 clinicians that report TUS/US findings apart from the PhD student. This can give high interobserver variability.

Apart from those, the mortality rate is high in F-ILD patients and will be expected high dropout rate. Therefore, the investigators are expecting to include patients according to our sample size calculation (34-117 patients).

Finally, the LORD study will contribute with knowledge on innovative methods to identification and prediction of F-ILD development over time due the study's follow-up design. Investigating a combination of different TUS/US modalities as single or composite markers of F-ILD disease dynamics is original and not previously conformed for this disease category. The observations from this study will not only fill out the existing knowledge gap, but also be able to point-out which future TUS/US markers to be used in order determine F-ILD disease severity, and thus be clinical implementable.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over 18 years.
* Diagnosis of IPF obtained on a multidisciplinary team conference .
* Diagnosis of PPF according to 2022 ATS/ERS/JRS/ALAT Clinical Practice Guideline.
* Ability for subject to comply with the requirements of the study.
* Informed consent.

Exclusion Criteria:

* Patients not willing to or able to give informed consent.
* Acute exacerbation in F-ILD < 4 weeks.
* Pregnant and breastfeeding mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from South Danish Center for ILD (SCILS) under the Department of Respiratory Medicine at Odense University Hospital, Denmark. SCILS receive patients suspected for ILD from both the primary sector within their local areas as well as from all other hospital departments within the region. Annually SCILS asses approximate 1.500 outpatient clinic patients, and 400 new patients referred for assessment.
  Respiratory physician that work in SCILS informed eligible patients regarding project and the PhD student contact them afterwards.
Sampling Method: Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Thoracic ultrasound/ ultrasound (TUS/US) measurments over 12 months in patients with F-ILD. | 12 months. The investigator group will examine patients in baseline (Day 0), after 6 months (day 180) and after 12 months (day 365).
  The investigators want to examine that TUS/US modalities such as B line artifacts (BLA) , interstitial syndrom (IS), pleural abnormalities (PA), diapgragm excursion (DE), lung ultarsound share wave elastography (LUSWE), appendicular lean mass (ALM) are clinically valuable, both individually and in combination for identifying F-ILD and monitoring disease activity.
  These modalities are expected to predict FVC (%), diffusion capacity of the lung for carbon monoxide (DLCO%), HRCT findings, and clinical symptoms.
  The invstigators hypothized that F-ILD patients with severe disease are present increased number of BLAs( more than 10 B-lines in minimum 2 lung zones), increased pleural irregularities (in milimeters), decreased DE (DE in milimeters), higher LUSWE velocities (meters and second to m/s), and lower ALM values (Kilogram and meters combined to report ALM kg/m2).
  The investigators wan to further these modalities serve as dynamic indicators of F-ILD disease activity over time.

SECONDARY OUTCOMES:
Measure the association and variability and observer variabilty. | 12 months. The investigator group will examine patients in baseline (Day 0), after 6 months (day 180) and after 12 months (day 365).
  Apart from the primary outcomes the investigator gruop wnat to asses the changes in TUS/US modalities with the HRCT Warrick score in the basline and after 365 days. According to our protocol all the included patients will examined with HRCT on baseline and after 365 days. So the investigators want to asses the association between HRCT severity by Warrick score ( a scale with the score from 0-30) with TUS/US changes.
  Furthermore the investigatores will plan to asses the intra- and inter- observational variability of TUS/US modalities. Only the PhD student is conductiing all the TUS/US scannings. Therefor it is necessary to exmine intra- and inter-obeservational variabilty.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper R Davidsen, MD,PhD, Principal Investigator — Department of Respiratory Medicine, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Man MA, Dantes E, Domokos Hancu B, Bondor CI, Ruscovan A, Parau A, Motoc NS, Marc M. Correlation between Transthoracic Lung Ultrasound Score and HRCT Features in Patients with Interstitial Lung Diseases. J Clin Med. 2019 Aug 11;8(8):1199. doi: 10.3390/jcm8081199. PMID 31405211
- [Background] Sperandeo M, Varriale A, Sperandeo G, Filabozzi P, Piattelli ML, Carnevale V, Decuzzi M, Vendemiale G. Transthoracic ultrasound in the evaluation of pulmonary fibrosis: our experience. Ultrasound Med Biol. 2009 May;35(5):723-9. doi: 10.1016/j.ultrasmedbio.2008.10.009. Epub 2008 Dec 27. PMID 19111972
- [Background] Safai Zadeh E, Gorg C, Prosch H, Kifjak D, Dietrich CF, Laursen CB, Findeisen H. Lung Ultrasound and Pleural Artifacts: A Pictorial Review. Diagnostics (Basel). 2024 Jan 13;14(2):179. doi: 10.3390/diagnostics14020179. PMID 38248056
- [Background] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905
- [Background] Clay R, Bartholmai BJ, Zhou B, Karwoski R, Peikert T, Osborn T, Rajagopalan S, Kalra S, Zhang X. Assessment of Interstitial Lung Disease Using Lung Ultrasound Surface Wave Elastography: A Novel Technique With Clinicoradiologic Correlates. J Thorac Imaging. 2019 Sep;34(5):313-319. doi: 10.1097/RTI.0000000000000334. PMID 29877916
- [Background] Zhang X, Zhou B, Osborn T, Bartholmai B, Kalra S. Lung Ultrasound Surface Wave Elastography for Assessing Interstitial Lung Disease. IEEE Trans Biomed Eng. 2019 May;66(5):1346-1352. doi: 10.1109/TBME.2018.2872907. Epub 2018 Oct 1. PMID 30281430
- [Background] Skaarup SH, Lokke A, Laursen CB. The Area method: a new method for ultrasound assessment of diaphragmatic movement. Crit Ultrasound J. 2018 Jun 27;10(1):15. doi: 10.1186/s13089-018-0092-5. PMID 29946769
- [Background] Mendoza L, Gogali A, Shrikrishna D, Cavada G, Kemp SV, Natanek SA, Jackson AS, Polkey MI, Wells AU, Hopkinson NS. Quadriceps strength and endurance in fibrotic idiopathic interstitial pneumonia. Respirology. 2014 Jan;19(1):138-43. doi: 10.1111/resp.12181. PMID 24033388
- [Background] du Bois RM, Albera C, Bradford WZ, Costabel U, Leff JA, Noble PW, Sahn SA, Valeyre D, Weycker D, King TE Jr. 6-Minute walk distance is an independent predictor of mortality in patients with idiopathic pulmonary fibrosis. Eur Respir J. 2014 May;43(5):1421-9. doi: 10.1183/09031936.00131813. Epub 2013 Dec 5. PMID 24311766
- [Background] Zhang X, Zhou B, Bartholmai B, Kalra S, Osborn T. A quantitative method for measuring the changes of lung surface wave speed for assessing disease progression of interstitial lung disease. Ultrasound Med Biol. 2019 Mar;45(3):741-748. doi: 10.1016/j.ultrasmedbio.2018.11.003. Epub 2018 Dec 29. PMID 30598191
- [Background] Zhang X, Osborn T, Zhou B, Meixner D, Kinnick RR, Bartholmai B, Greenleaf JF, Kalra S. Lung Ultrasound Surface Wave Elastography: A Pilot Clinical Study. IEEE Trans Ultrason Ferroelectr Freq Control. 2017 Sep;64(9):1298-1304. doi: 10.1109/TUFFC.2017.2707981. PMID 28866480
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753
- [Background] Davidsen JR, Schultz HHL, Henriksen DP, Iversen M, Kalhauge A, Carlsen J, Perch M, Graumann O, Laursen CB. Lung Ultrasound in the Assessment of Pulmonary Complications After Lung Transplantation. Ultraschall Med. 2020 Apr;41(2):148-156. doi: 10.1055/a-0783-2466. Epub 2018 Nov 9. PMID 30414162
- [Background] Laursen CB, Clive A, Hallifax R, Pietersen PI, Asciak R, Davidsen JR, Bhatnagar R, Bedawi EO, Jacobsen N, Coleman C, Edey A, Via G, Volpicelli G, Massard G, Raimondi F, Evison M, Konge L, Annema J, Rahman NM, Maskell N. European Respiratory Society statement on thoracic ultrasound. Eur Respir J. 2021 Mar 4;57(3):2001519. doi: 10.1183/13993003.01519-2020. Print 2021 Mar. PMID 33033148
- [Background] Osterwalder J, Polyzogopoulou E, Hoffmann B. Point-of-Care Ultrasound-History, Current and Evolving Clinical Concepts in Emergency Medicine. Medicina (Kaunas). 2023 Dec 15;59(12):2179. doi: 10.3390/medicina59122179. PMID 38138282
- [Background] Sofiudottir BK, Harders S, Laursen CB, Lage-Hansen PR, Nielsen SM, Just SA, Christensen R, Davidsen JR, Ellingsen T. Detection of Interstitial Lung Disease in Rheumatoid Arthritis by Thoracic Ultrasound: A Diagnostic Test Accuracy Study. Arthritis Care Res (Hoboken). 2024 Sep;76(9):1294-1302. doi: 10.1002/acr.25351. Epub 2024 Jun 23. PMID 38622106
- [Background] Otaola M, Paulin F, Rosemffet M, Balcazar J, Perandones M, Orausclio P, Cazenave T, Rossi S, Marciano S, Schneeberger E, Citera G. Lung ultrasound is a promising screening tool to rule out interstitial lung disease in patients with rheumatoid arthritis. Respirology. 2024 Jul;29(7):588-595. doi: 10.1111/resp.14679. Epub 2024 Feb 18. PMID 38369685
- [Background] Flaherty KR, Wells AU, Cottin V, Devaraj A, Walsh SLF, Inoue Y, Richeldi L, Kolb M, Tetzlaff K, Stowasser S, Coeck C, Clerisme-Beaty E, Rosenstock B, Quaresma M, Haeufel T, Goeldner RG, Schlenker-Herceg R, Brown KK; INBUILD Trial Investigators. Nintedanib in Progressive Fibrosing Interstitial Lung Diseases. N Engl J Med. 2019 Oct 31;381(18):1718-1727. doi: 10.1056/NEJMoa1908681. Epub 2019 Sep 29. PMID 31566307
- [Background] Raghu G, Remy-Jardin M, Richeldi L, Thomson CC, Inoue Y, Johkoh T, Kreuter M, Lynch DA, Maher TM, Martinez FJ, Molina-Molina M, Myers JL, Nicholson AG, Ryerson CJ, Strek ME, Troy LK, Wijsenbeek M, Mammen MJ, Hossain T, Bissell BD, Herman DD, Hon SM, Kheir F, Khor YH, Macrea M, Antoniou KM, Bouros D, Buendia-Roldan I, Caro F, Crestani B, Ho L, Morisset J, Olson AL, Podolanczuk A, Poletti V, Selman M, Ewing T, Jones S, Knight SL, Ghazipura M, Wilson KC. Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline. Am J Respir Crit Care Med. 2022 May 1;205(9):e18-e47. doi: 10.1164/rccm.202202-0399ST. PMID 35486072
- [Background] Cottin V, Hirani NA, Hotchkin DL, Nambiar AM, Ogura T, Otaola M, Skowasch D, Park JS, Poonyagariyagorn HK, Wuyts W, Wells AU. Presentation, diagnosis and clinical course of the spectrum of progressive-fibrosing interstitial lung diseases. Eur Respir Rev. 2018 Dec 21;27(150):180076. doi: 10.1183/16000617.0076-2018. Print 2018 Dec 31. PMID 30578335
- [Background] Hoyer N, Prior TS, Bendstrup E, Wilcke T, Shaker SB. Risk factors for diagnostic delay in idiopathic pulmonary fibrosis. Respir Res. 2019 May 24;20(1):103. doi: 10.1186/s12931-019-1076-0. PMID 31126287
- [Background] Pinal-Fernandez I, Pallisa-Nunez E, Selva-O'Callaghan A, Castella-Fierro E, Simeon-Aznar CP, Fonollosa-Pla V, Vilardell-Tarres M. Pleural irregularity, a new ultrasound sign for the study of interstitial lung disease in systemic sclerosis and antisynthetase syndrome. Clin Exp Rheumatol. 2015 Jul-Aug;33(4 Suppl 91):S136-41. Epub 2015 Aug 27. PMID 26315813
- [Background] Bujang MA, Adnan TH. Requirements for Minimum Sample Size for Sensitivity and Specificity Analysis. J Clin Diagn Res. 2016 Oct;10(10):YE01-YE06. doi: 10.7860/JCDR/2016/18129.8744. Epub 2016 Oct 1. PMID 27891446
- [Background] Simpson T, Barratt SL, Beirne P, Chaudhuri N, Crawshaw A, Crowley LE, Fletcher S, Gibbons MA, Hallchurch P, Horgan L, Jakaityte I, Lewis T, McLellan T, Myall KJ, Miller R, Smith DJF, Stanel S, Thillai M, Thompson F, Wallis T, Wu Z, Molyneaux PL, West AG. The burden of progressive fibrotic interstitial lung disease across the UK. Eur Respir J. 2021 Jul 8;58(1):2100221. doi: 10.1183/13993003.00221-2021. Print 2021 Jul. PMID 33678609
- [Background] Wijsenbeek M, Kreuter M, Olson A, Fischer A, Bendstrup E, Wells CD, Denton CP, Mounir B, Zouad-Lejour L, Quaresma M, Cottin V. Progressive fibrosing interstitial lung diseases: current practice in diagnosis and management. Curr Med Res Opin. 2019 Nov;35(11):2015-2024. doi: 10.1080/03007995.2019.1647040. Epub 2019 Aug 2. PMID 31328965
- [Background] Laursen CB, Sloth E, Lassen AT, Davidsen JR, Lambrechtsen J, Henriksen DP, Madsen PH, Rasmussen F. Does point-of-care ultrasonography cause discomfort in patients admitted with respiratory symptoms? Scand J Trauma Resusc Emerg Med. 2015 Jun 13;23:46. doi: 10.1186/s13049-015-0127-x. PMID 26071404
- [Background] Mohammad Reza Beigi D, Pellegrino G, Loconte M, Landini N, Mattone M, Paone G, Truglia S, Di Ciommo FR, Bisconti I, Cadar M, Stefanantoni K, Panebianco V, Conti F, Riccieri V. Lung ultrasound compared to computed tomography detection and automated quantification of systemic sclerosis-associated interstitial lung disease: preliminary study. Rheumatology (Oxford). 2024 May 2;63(5):1240-1245. doi: 10.1093/rheumatology/kead324. PMID 37399086
- [Background] Di Carlo M, Tardella M, Filippucci E, Carotti M, Salaffi F. Lung ultrasound in patients with rheumatoid arthritis: definition of significant interstitial lung disease. Clin Exp Rheumatol. 2022 Mar;40(3):495-500. doi: 10.55563/clinexprheumatol/gioptt. Epub 2021 Apr 23. PMID 33938789
- [Background] Manolescu D, Oancea C, Timar B, Traila D, Malita D, Birsasteanu F, Tudorache V. Ultrasound mapping of lung changes in idiopathic pulmonary fibrosis. Clin Respir J. 2020 Jan;14(1):54-63. doi: 10.1111/crj.13101. Epub 2019 Nov 14. PMID 31675455
- [Background] Manolescu D, Davidescu L, Traila D, Oancea C, Tudorache V. The reliability of lung ultrasound in assessment of idiopathic pulmonary fibrosis. Clin Interv Aging. 2018 Mar 22;13:437-449. doi: 10.2147/CIA.S156615. eCollection 2018. PMID 29606857
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Prado-Costa R, Rebelo J, Monteiro-Barroso J, Preto AS. Ultrasound elastography: compression elastography and shear-wave elastography in the assessment of tendon injury. Insights Imaging. 2018 Oct;9(5):791-814. doi: 10.1007/s13244-018-0642-1. Epub 2018 Aug 17. PMID 30120723
- [Background] Santana PV, Prina E, Albuquerque AL, Carvalho CR, Caruso P. Identifying decreased diaphragmatic mobility and diaphragm thickening in interstitial lung disease: the utility of ultrasound imaging. J Bras Pneumol. 2016 Apr;42(2):88-94. doi: 10.1590/S1806-37562015000000266. PMID 27167428
- [Background] Boccatonda A, Decorato V, Cocco G, Marinari S, Schiavone C. Ultrasound evaluation of diaphragmatic mobility in patients with idiopathic lung fibrosis: a pilot study. Multidiscip Respir Med. 2018 Dec 14;14:1. doi: 10.1186/s40248-018-0159-y. eCollection 2019. PMID 30651988
- [Background] Hasan AA, Makhlouf HA. B-lines: Transthoracic chest ultrasound signs useful in assessment of interstitial lung diseases. Ann Thorac Med. 2014 Apr;9(2):99-103. doi: 10.4103/1817-1737.128856. PMID 24791173
- [Background] Tardella M, Di Carlo M, Carotti M, Filippucci E, Grassi W, Salaffi F. Ultrasound B-lines in the evaluation of interstitial lung disease in patients with systemic sclerosis: Cut-off point definition for the presence of significant pulmonary fibrosis. Medicine (Baltimore). 2018 May;97(18):e0566. doi: 10.1097/MD.0000000000010566. PMID 29718851
- [Background] Warrick JH, Bhalla M, Schabel SI, Silver RM. High resolution computed tomography in early scleroderma lung disease. J Rheumatol. 1991 Oct;18(10):1520-8. PMID 1765976
- [Background] Poosiri S, Krisanachinda A, Khamwan K. Evaluation of patient radiation dose and risk of cancer from CT examinations. Radiol Phys Technol. 2024 Mar;17(1):176-185. doi: 10.1007/s12194-023-00763-w. Epub 2023 Dec 4. PMID 38048023
- [Background] Lederer C, Storman M, Tarnoki AD, Tarnoki DL, Margaritopoulos GA, Prosch H. Imaging in the diagnosis and management of fibrosing interstitial lung diseases. Breathe (Sheff). 2024 Mar;20(1):240006. doi: 10.1183/20734735.0006-2024. Epub 2024 May 14. PMID 38746908
- [Background] Wijsenbeek M, Cottin V. Spectrum of Fibrotic Lung Diseases. Reply. N Engl J Med. 2020 Dec 17;383(25):2485-2486. doi: 10.1056/NEJMc2031135. No abstract available. PMID 33326734